CLINICAL TRIAL: NCT03707522
Title: The Effect of Growth Mindset Psychoeducation on Modifiable Risk Factors for Common Mental Disorders
Brief Title: Growth Mindset Psychoeducation for Modifiable Risk Factors for CMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Principal Investigator, Martha Zimmermann, Principal Investigator, University of Nevada, Reno
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: Psychoeducation for CMD
Record Dates: First submitted 2018-10-09; First posted 2018-10-16 (Actual); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Growth mindset + MRF Information (Experimental): Online growth mindset interactive article followed by equal length interactive article describing the relationship between modifiable risk factors (MRF) and mental health outcomes
  Interventions: Behavioral: Growth mindset; Behavioral: Modifiable risk factor (MRF) information
- Control + MRF information (Experimental): Online daily activity scheduling interactive article (control) followed by equal length interactive article describing the relationship between modifiable risk factors and mental health outcomes
  Interventions: Behavioral: Modifiable risk factor (MRF) information; Behavioral: Control
- Control + Growth mindset (Experimental): Online growth mindset interactive article followed by equal length online daily activity scheduling interactive article (control)
  Interventions: Behavioral: Growth mindset; Behavioral: Control
- Control + Control (Placebo Comparator): 2 doses online daily activity scheduling interactive article (control)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Growth mindset — 10 minute interactive article describing neuroplasticity
  Arms: Control + Growth mindset; Growth mindset + MRF Information
Behavioral: Modifiable risk factor (MRF) information — 10 minute interactive article describing modifiable risk factors for depression and anxiety
  Arms: Control + MRF information; Growth mindset + MRF Information
Behavioral: Control — 10 minute interactive article describing activity scheduling
  Arms: Control + Control; Control + Growth mindset; Control + MRF information

SUMMARY:
The present study aims to determine the effect of presenting psychoeducation emphasizing "growth-mindset," and information on modifiable risk factors (e.g., social contact, physical activity) on engagement with modifiable risk factors. The investigators hypothesize that psychoeducation emphasizing that mental health is malleable will increase the participant's engagement with risk factors outlined in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* College freshmen

Exclusion Criteria:

* Not fluent in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Papa, PhD, Principal Investigator — University of Nevada, Reno
Locations (1):
- University of Nevada, Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lee JP, Lee RM, Hu AW, Kim OM. Ethnic Identity as a Moderator against Discrimination for Transracially and Transnationally Adopted Korean American Adolescents. Asian Am J Psychol. 2015 Jun;6(2):154-163. doi: 10.1037/a0038360. PMID 26273427
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Zazpe I, Bes-Rastrollo M, Ruiz-Canela M, Sanchez-Villegas A, Serrano-Martinez M, Martinez-Gonzalez MA. A brief assessment of eating habits and weight gain in a Mediterranean cohort. Br J Nutr. 2011 Mar;105(5):765-75. doi: 10.1017/S0007114510004149. Epub 2010 Dec 8. PMID 21138604
- [Background] Ottenbreit ND, Dobson KS. Avoidance and depression: the construction of the cognitive-behavioral avoidance scale. Behav Res Ther. 2004 Mar;42(3):293-313. doi: 10.1016/S0005-7967(03)00140-2. PMID 14975771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: College students recruited via e-mail
Period: Overall Study
Arm/Group | Growth Mindset + MRF Information | Control + MRF Information | Control + Growth Mindset | Control + Control
Started | 31 | 36 | 52 | 43
Completed | 7 | 9 | 11 | 7
Not Completed | 24 | 27 | 41 | 36
Not completed — Lost to Follow-up | 24 | 27 | 41 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Growth Mindset + MRF Information | Control + MRF Information | Control + Growth Mindset | Control + Control | Total
Number analyzed (Participants) | 31 | 36 | 52 | 43 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.06 (.25) | 18.00 (.00) | 18.02 (.14) | 18.07 (.26) | 18.04 (.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 11 | 14 | 43
  Male | 24 | 25 | 41 | 29 | 119
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnciity: White | 17 | 22 | 29 | 27 | 95
  Race/ethnciity: Hispanic or Latino | 5 | 5 | 6 | 8 | 24
  Race/ethnciity: Black or African-American | 1 | 1 | 3 | 0 | 5
  Race/ethnciity: Native American or American Indian | 0 | 2 | 1 | 0 | 3
  Race/ethnciity: Asian/Pacific Islander | 4 | 5 | 9 | 5 | 23
  Race/ethnciity: Other | 4 | 1 | 4 | 3 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 36 | 52 | 43 | 162
PHQ-9 (Depression severity) [Mean (Standard Deviation); unit: units on a scale] — Severity of depression was be measured via the Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001), a 9-item questionnaire associated containing one item for each symptom of MDD as specified by the DSM. Scores range from 0-27. Scores 0-4 indicate minimal depression, 5-9 indicate mild depression, 10-14 moderate depression, 15-19 moderately severe depression, 20-27 severe depression.
  units on a scale | 7.06 (6.01) | 5.28 (5.22) | 5.62 (5.34) | 9.65 (7.93) | 6.89 (6.43)
GAD-7 (Anxiety severity) [Mean (Standard Deviation); unit: units on a scale] — Anxiety severity was measured using the Generalized Anxiety Disorder 7-item scale (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006). The GAD-7 is a common, brief measure of anxiety symptom severity (α = .92). The range of scores is from 0-21. A score of 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates severe anxiety.
  units on a scale | 5.97 (5.31) | 5.25 (5.82) | 5.52 (5.08) | 8.26 (6.53) | 6.27 (5.78)

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer & Williams, 2001)
Description: 9-item questionnaire associated containing one item for each symptom of MDD as specified by the DSM. Items consist of a 4-point Likert scale (0="Not at all" to 3="Nearly every day"). Minimum score is 0, maximum score is 27. Higher scores indicate greater depression severity.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Growth Mindset + MRF Information | Control + MRF Information | Control + Growth Mindset | Control + Control
Number analyzed (Participants) | 7 | 9 | 11 | 7
units on a scale | 5.50 (7.34) | 4.57 (3.15) | 6.70 (3.37) | 13.14 (7.52)

2. Primary Outcome: Generalized Anxiety Disorder-7 (GAD-7; Spitzer, Kroenke, Williams & Lowe, 2006)
Description: 7-item scale, common, brief measure of anxiety symptom severity. Items consist of a 4-point Likert scale (0="Not at all" to 3="Nearly every day"). Minimum score is 0, maximum score is 21. Higher scores indicate greater anxiety symptom severity.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Growth Mindset + MRF Information | Control + MRF Information | Control + Growth Mindset | Control + Control
Number analyzed (Participants) | 6 | 7 | 10 | 7
units on a scale | 3.67 (5.75) | 4.43 (6.29) | 6.90 (4.68) | 12.14 (7.69)

3. Secondary Outcome: Cognitive and Behavioral Avoidance Scale (CBAS, Ottenbreit & Dobson, 2003)
Description: The scale contains 31 items assessing cognitive avoidance and behavioral avoidance of social and non-social avoidance. The scale uses a 5-item Likert scale (1="Not at all true for me" to 5="Extremely true for me"). Total scale range from 0-155. The behavioral social factor contains 8 items. Items are summed. Minimum score is 8, maximum score is 40. The cognitive nonsocial scale contains 10 items. Minimum score is 10. Maximum score is 50. The cognitive social subscale consists of 7 items. Minimum score is 7, maximum score is 35. The behavioral nonsocial subscale consists of 6 items. Minimum score is 6, maximum score is 30. Higher scores indicate higher levels of avoidance.
Time Frame: 3 months
Population: 1 participant completed primary but not secondary outcome measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Growth Mindset + MRF Information | Control + MRF Information | Control + Growth Mindset | Control + Control
Number analyzed (Participants) | 7 | 9 | 10 | 7
units on a scale | 52.1 (19.6) | 57.3 (22.9) | 54.8 (17.8) | 74.3 (25.2)

4. Secondary Outcome: Substance Use Measure (Lee et al., 2015)
Description: 3-item substance use measure including frequency of alcohol use, cigarette use and drug use. Items are measured using a five-point Likert scale (1="never or not at all" to 5="almost always"). The scale is scored by summing items. Minimum score is 3, maximum score is 15. Higher scores indicate more frequent substance use.
Time Frame: 3 months
Population: 2 participants completed primary but not secondary outcomes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Growth Mindset + MRF Information | Control + MRF Information | Control + Growth Mindset | Control + Control
Number analyzed (Participants) | 7 | 9 | 9 | 7
units on a scale | 3.9 (1.5) | 3.2 (.7) | 3.6 (1.3) | 4.9 (2.5)

5. Secondary Outcome: Positive Reframing; Brief COPE (B-COPE; Carver, 1997)
Description: 28-item scale assessing various dimensions of healthy and unhealthy coping. This include 14 subscales: self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion, and self-blame. Each subscale consists of two items. Subscales are scored by summing items. Scale consists of 4-item Likert scale (1="I haven't been doing this at all" to 4 "I've been doing this a lot"). Minimum score is 2, maximum score is 8 on each subscale. Higher scores indicate greater use of coping strategy. Positive reframing subscale was used.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Growth Mindset + MRF Information | Control + MRF Information | Control + Growth Mindset | Control + Control
Number analyzed (Participants) | 7 | 9 | 11 | 7
units on a scale | 2.9 (1.1) | 2.9 (1.1) | 2.4 (.83) | 3.2 (1.0)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Growth Mindset + MRF Information | Control + MRF Information | Control + Growth Mindset | Control + Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT03707522/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT03707522/ICF_001.pdf